CLINICAL TRIAL: NCT04653038
Title: An Open-label, Multi-cohort, Multi-center Phase I Study Evaluating the Efficacy and Safety of MGD013 in Patients With Unresectable, Recurrent or Metastatic Malignant Melanoma
Brief Title: A Study to Evaluate the Safety and Efficacy of MGD013 in Patients With Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: rapid changes in the treatment mode of melanoma worldwide and in China and the development strategy change
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZL-1301-003
Record Dates: First submitted 2020-11-16; First posted 2020-12-04 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Unresectable, Recurrent or Metastatic Melanoma; Untreated Mucosal or Acral Lentiginous Melanoma
Keywords: Melanoma; MGD013
MeSH Terms: conditions — Recurrence; Melanoma

STUDY DESIGN:
Intervention Model Description: ① Cohort 1: patients with unresectable, recurrent or metastatic melanoma who have failed prior immune checkpoint inhibitor therapy; ② Cohort 2: patients with untreated, unresectable recurrent or metastatic, mucosal or acral lentiginous melanoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Unresectable, recurrent or metastatic melanoma (Experimental): Cohort1: patients with unresectable, recurrent or metastatic melanoma who have failed prior immune checkpoint inhibitor therapy
  Interventions: Drug: MGD013
- Untreated mucosal or acral lentiginous melanoma (Experimental): Cohort2: patients with untreated, unresectable recurrent or metastatic, mucosal or acral lentiginous melanoma
  Interventions: Drug: MGD013

INTERVENTIONS:
Drug: MGD013 — A fixed dose of MGD013 600mg IV Q2W will be administered to subjects

SUMMARY:
This is an open-label, multi-cohort, multi-center Phase I clinical trial to evaluate the efficacy and safety of MGD013 in ① Cohort 1: patients with unresectable, recurrent or metastatic melanoma who have failed prior immune checkpoint inhibitor therapy; ② Cohort 2: patients with untreated, unresectable recurrent or metastatic, mucosal or acral lentiginous melanoma.

DETAILED DESCRIPTION:
The study is conducted in two parts for both Cohort 1 and Cohort 2. Part I: Safety evaluation and efficacy exploration for MGD013. Part II: Efficacy expansion based on results from Part I to further evaluate the efficacy effect of MGD013.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary and able to provide signed informed consent form
* Male or female aged ≥ 18 years
* Patient can comply with protocol requirements as assessed by the investigator
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, or 1
* Histologically confirmed unresectable recurrent or metastatic melanoma:

  * Cohort 1: The pathological type is cutaneous or acral lentiginous, or unknown origin. Progressive or recurrent disease on at least one prior line of systemic therapies. In addition, prior systemic therapies must include one line of anti-PD-(L)1 and/or anti-CTLA-4 immune checkpoint inhibitors. Patients with BRAF-mutated or KIT-mutated/amplified melanoma, and prior treatment with vemurafenib or imatinib is not mandatory;
  * Cohort 2: Histologically confirmed pathological type is acral lentiginous or mucosal. No prior systemic therapy for recurrent or metastatic disease.
* Patients with at least one measurable lesion according to irRECIST; assessed by investigator per irRECIST criteria to establish a baseline tumor assessment, and should be performed within 28 days prior to the first dose.

Exclusion Criteria:

* The pathological type of patient is:

  * Cohort 1: Mucosal melanoma; uveal melanoma;
  * Cohort 2: Cutaneous melanoma; uveal melanoma; melanoma of unknown origin; known BRAF mutation or KIT mutation/amplification.
* Central nervous system metastases with clinical symptoms. Patients with prior central nervous system metastases who have received local therapy, have stable disease for ≥ 4 weeks, and meet the following criteria can be enrolled:

  * No treatment for central nervous system metastases during the screening period (e.g., surgery, radiotherapy, mannitol, corticosteroid therapy-prednisolone > 10 mg per day or equivalent dose)
  * No progression of central nervous system lesions on MRI or CT within 14 days prior to start of study treatment
  * No meningeal metastasis or notochord compression
* Subjects with a history of symptomatic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired pulmonary function or may interfere with the detection and treatment of suspected drug-related pulmonary adverse reactions;
* Prior treatment with any antibody/drug targeting the regulation of T cell function (immune checkpoint) (e.g., anti-LAG-3, anti-0X-40, anti-CD137, anti-TIM-3, anti-TIGIT, IDO)
* Patients who have previously received immune checkpoint inhibitors (e.g., anti-PD-(L)1, anti-CTLA-4 antibody) are not included if they experience any of the following immune checkpoint-related adverse events, regardless of recovery:

  * ≥ Grade 3 ocular adverse events
  * Grade 4 liver function abnormalities
  * Grade ≥ 3 neurologic adverse reactions
  * ≥ Grade 3 colitis
  * ≥ Grade 3 renal adverse reactions
  * ≥ Grade 3 pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 12 months after dosed
  Objective Response Rate (ORR) is defined as the proportion of patients with a best response of CR or PR in enrolled patients, which is assessed by Independent Review Committee (IRC) per RECIST v1.1

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 12 months after dosed
  Objective Response Rate (ORR) as assessed by Investigator per RECIST v1.1
Objective Response Rate (ORR) | Approximately 12 months after dosed
  Objective Response Rate (ORR) as assessed by Investigator and IRC per irRECIST.
Overall Survival (OS) | Approximately 24 months
  Overall Survival (OS) is defined as the time from patient enrollment to death due to any cause
Progression-free Survival (PFS) | Approximately 12 months after dosed
  Progression-free Survival (PFS) is defined as the time from patient enrollment to tumor progression or death due to any cause. Progression is assessed per RECIST 1.1 and irRECIST criteria, respectively
Disease Control Rate (DCR) | Approximately 12 months after dosed
  Disease Control Rate (DCR) is defined as the time from patient enrollment to tumor progression or death due to any cause. The tumor progression is assessed per RECIST 1.1 and irRECIST criteria, respectively
Duration of Response (DoR) | Approximately 12 months after dosed
  Duration of Response (DoR) is defined as the time from radiographic response to disease progression or death in patients with a best response of CR or PR, assessed per RECIST 1.1 and irRECIST criteria, respectively
Survival Rate | Approximately 12 months after dosed
  Survival Rate is defined as the proportion of surviving patients at the corresponding time point. Survival rates at 6 and 12 months will be analyzed in this study
Incidence of Abnormal Laboratory value | Approximately 24 months
  Incidence of abnormal laboratory is defined as the proportion of patients who have abnormal laboratory value not prior to the initiation of MGD013 administration
Incidence of Adverse Events | Approximately 24 months
  The incidence of adverse events is defined as the proportion of the patients who have adverse event(s) enrolled in this study.
Incidence of Treatment-Emergent Adverse Events | Approximately 24 months.
  The incidence of treatment-emergent adverse event is defined as any event not present prior to the initiation of MGD013 treatment or any event already present that worsens in either intensity or frequency following exposure to MGD013 administration.
Maximum Serum Concentration (Cmax) | Approximately 3 months.
  The maximum serum concentration (Cmax, ng/ml) is defined as the maximum (or peak) serum concentration that MGD013 achieves in patients after the MGD013 administration at a corresponding timepoint.
Trough Serum Concentration (Ctrough) | Approximately 3 months
  The through serum concentration (Cmin, ng/ml) is defined as the minimum (or through) serum concentration reached by MGD013 prior to administration of a second dose.
Immunogenicity of MGD013 | Approximately 6 months after dosed
  Immunogenicity is defined as the positivity measured as the anti-MGD013 antibody induced in serum after MGD013 is administrated into human body at corresponding timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Jun GUO, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (13):
- China (13):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Xi’an, Shanxi
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Sir Run Shaw Hospital, School Of Medicine ,Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang